CLINICAL TRIAL: NCT05117450
Title: Comparison of HYDROLINK™ and HeprAN™ mEmbranes in a Per Dialytic Heparin Weaning Strategy in Chronic Hemodialysis Patients
Acronym: RESTIT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PO20179*
Record Dates: First submitted 2021-08-06; First posted 2021-11-11 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Renal Insufficiency
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HeprAN first (Active Comparator): Each included patient will have hemodialysis sessions with HeprAN membrane and then HYDROLINK
  Interventions: Device: Decrease per-dialytic heparin therapy
- HYDROLINK first (Active Comparator): Each included patient will have hemodialysis sessions with HYDROLINK and then HeprAN membrane
  Interventions: Device: Decrease per-dialytic heparin therapy

INTERVENTIONS:
Device: Decrease per-dialytic heparin therapy — Decrease per-dialytic heparin therapy with the HYDROLINK membrane (dialyzer NV-21U, surface 2.1m², Toray industry, Tokyo, Japan) and with the HeprAN membrane (dialyzer Evodial 2.2, surface 2.15 m2, Hospal SAS, Meyzieu, France)

SUMMARY:
Chronic kidney disease (CKD) results from the progressive and irreversible destruction of the kidneys. As of December 31, 2018, there were 89,692 people in France undergoing replacement therapy, including 49,271 (55%) on dialysis and 40,421 (45%) with a functioning kidney transplant. The primary treatment modality is currently hemodialysis. It is known to activate the coagulation cascade and blood platelets, leading to thrombus formation and premature termination of the hemodialysis session. This loss of circuitry results in a decrease in session time leading to an insufficient dialysis dose and blood loss in patients who are already often anemic due to their chronic renal failure.

To avoid this complication, current recommendations recommend the use of unfractionated heparin (UFH) or low molecular weight heparin (LMWH) during the hemodialysis session at the cost of an obligatory hemorrhagic risk due to the systemic administration of heparin. However, this risk of bleeding is already very high, due to platelet dysfunction, a direct consequence of uremic toxin impregnation in these patients. In addition, this hemodialysis population is frequently exposed to antiplatelet agents and anticoagulants (heparin or VKA), which aggravate the hemorrhagic risk inherent to renal pathology.

In this context, bioactive membranes such as the HeprAN™ membrane, coated in heparin, have been developed to minimize or even eliminate the need for anticoagulation during sessions in chronic hemodialysis patients. Several studies with this membrane have demonstrated the absence of the need for additional heparin in populations with no particular bleeding risk and in populations at risk of bleeding: post-operative (HepZero study), patients on VKA.

The HYDROLINK™ membrane offers the same anticoagulant prospects as the HeprAN™ membrane, but its mode of action involves the use of a copolymer with hydrophilic properties, making it possible to avoid the presence of heparin. This membrane would have an influence on platelet aggregation. It would also make it possible to avoid the risk of heparin-induced thrombocytopenia (HIT) by completely excluding heparin from the dialysis session

DETAILED DESCRIPTION:
The aim of this study is to compare the HYDROLINK™ membrane to the HeprAN™ membrane in a large-scale trial with the strategy of minimizing the dose of peridialytic heparin in order to reduce the risk of bleeding in chronic hemodialysis patients.

Participation in the research will be offered at the time of a hemodialysis session to any eligible patient, i.e., over 18 years of age, who has been on chronic hemodialysis for at least 3 months at a rate of three times a week and who has given their consent to this study. A cross over trial will be performed. Each included patient will have hemodialysis sessions with HYDROLINK™ and HeprAN™ membrane.

ELIGIBILITY:
inclusion criteria :

* Patients with Age > 18 years
* Chronic hemodialysis for at least 3 months
* Hemodialysis three times a week
* On per dialytic heparin therapy (UFH or LMWH)
* Affiliated to the French Social Security
* Having given their consent for this study

exclusion criteria :

* Patients undergoing Hemodiafiltration (HDF)
* Pregnant or lactating woman
* Patient participating in another interventional study
* Persons deprived of liberty by judicial or administrative decision
* Adults under legal protection (under guardianship or curators)
* Persons under a legal protection measure
* Patients with a history of HIT
* Patients with acquired or congenital coagulation disorders
* Pathology with active neoplasia (Myeloma, Waldenström disease, solid cancers)
* Patient on an ACE inhibitor (ACE inhibitor)
* Patient requiring transfusion during the study period
* Patient not hemoglobin-stabilized (mean Hb < 10g/dL or >12 g/dL in the previous month)
* Patient septic or with significant inflammation (defined as C-reactive protein > 25mg/L) at the time of inclusion
* Patient requiring per-dialytic parenteral nutrition
* Patient requiring hospitalization or scheduled surgery during the study period
* Vascular access (Arteriovenous Fistula or Arteriovenous graft with the possibility of 2 needles) not allowing a sufficient blood pump flow (< 300 mL/min determined during the screening phase = blood flow prescribed by the nephrologist)
* Patient dialyzing on catheter ("single line" or "double line") or in unipuncture on Arteriovenous fistula on the day of the screening session
* Net ultrafiltration on the day of the screening session > 4000 mL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Estimated)
Dates: Start 2021-11-17 (Actual); Primary Completion 2026-11-17 (Estimated); Study Completion 2026-12-17 (Estimated)

PRIMARY OUTCOMES:
number of hemodialysis session success without heparin | 4 weeks
  The success of the hemodialysis session is defined by a dialysis time> 95% of the prescribed time

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, Reims, France

IPD SHARING:
Plan to Share IPD: Undecided